CLINICAL TRIAL: NCT01680354
Title: Comparative Study of Surgical Laser Correction of Astigmatism
Brief Title: Surgical Correction of Astigmatism
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Institution changed surgical method to small incision lenticule extraction. Study never started.
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anders Ivarsen, MD, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUH_ASTIGMATISM
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReLEx (Active Comparator): One eye is treated with ReLEx the other with LASIK
  Interventions: Procedure: ReLEx
- LASIK (Active Comparator): One eye is treated with ReLEx the other with LASIK
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: ReLEx
  Other Names: Device: Carl Zeiss Meditec Visumax Femtosecond Laser
  Arms: ReLEx
Procedure: LASIK
  Other Names: Device: Carl Zeiss Meditec MEL-80 excimer laser
  Arms: LASIK

SUMMARY:
Laser correction for myopia and astigmatism using an excimer laser has been performed with success for several years.

During the last 2 years, a new method for correction of refractive errors has emerged. In the method (ReLex) a femtosecond laser is used to cut a lenticule in the corneal stroma that is subsequently removed. For simple myopia this method has proved effective and on par with excimer baser LASIK. However, it remains to be determined if ReLEx is as effective in the treatment of astigmatism.

In the study, patients with high astigmatism are treated with conventional LASIK for astigmatism in one eye and with ReLEx for astigmatism in the other.

ELIGIBILITY:
Inclusion Criteria:

* Myopic astigmatism between -2.0 and -5.0 diopters
* Maximal difference in spherical equivalent refraction of 2 D between eyes
* No ocular or systemic disease
* Not pregnant or breastfeeding
* Minimum BSCVA of 0.8 (decimal)
* Normal corneal topography
* Sufficient corneal thickness to allow the treatment

Exclusion Criteria:

* Subjects not fulfilling the above criteria

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 year

SECONDARY OUTCOMES:
Refraction | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Aarhus University Hospital, Aarhus, Denmark